CLINICAL TRIAL: NCT01515553
Title: A Randomized, Double-blind, Single-centre, Two-period, Cross-over Trial in Healthy Subjects Investigating the Bioequivalence Between the Phase 3a Formulation of Liraglutide (Formulation 4) and the Planned Phase 3b Formulation (Final Formulation 4)
Brief Title: Bioequivalence of Two Liraglutide Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1692; 2006-004283-31 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation 4 (Experimental)
  Interventions: Drug: liraglutide
- Final formulation 4 (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Two single doses of 0.72 mg liraglutide administered subcutaneously on two different dosing occasions separated by a wash-out period

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to test for bioequivalence of the phase 3a formulation of liraglutide (formulation 4) and the liraglutide formulation planned for phase 3b trials (final formulation 4).

ELIGIBILITY:
Inclusion Criteria:

* Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs and blood and urinary laboratory assessments
* BMI (Body Mass Index) of 18.0-27.0 kg/m^2, both inclusive

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders that may interfere with the objectives of the trial, as judged by the Investigator
* Impaired renal function
* Any clinically significant abnormal ECG, as judged by the Investigator
* Active hepatitis B and/or active hepatitis C
* Positive human immunodeficiency virus (HIV) antibodies
* Known or suspected allergy to trial product(s) or related products
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
* History of alcoholism or drug abuse, or positive results in alcohol or drug screens
* Smoking of more than 5 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing (theophylline, caffeine or theobromine) beverages and foods (coffee, tea, soft drinks such as red bull, cola, chocolate) as judged by the Investigator
* Excessive consumption of a diet deviating from a normal diet as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (0-t)
Cmax, maximum concentration

SECONDARY OUTCOMES:
Area under the curve (0-infinity)
Relative bioavailability
Time to reach maximum (tmax)
Terminal elimination half life (t½)
Terminal elimination rate constant
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Lund, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com